CLINICAL TRIAL: NCT06543277
Title: Safety and Feasibility of Paired taVNS With Upper Limb Rehabilitation in Incomplete Spinal Cord Injury
Brief Title: Safety and Feasibility of Paired Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) With Upper Limb Rehabilitation in Incomplete Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Mission Connect (Unknown)
Responsible Party: Principal Investigator, Radha Korupolu, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-24-0346
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Chronic Incomplete Cervical Spinal Cord Injury (SCI)
Keywords: spinal cord injury (SCI); upper arm rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) (Experimental)
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Participants will receive 18 goal-directed upper extremity rehabilitation therapy sessions with paired taVNS over six weeks, followed by a 90-day home exercise program.

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of transcutaneous auricular Vagus Nerve Stimulation (taVNS) paired with upper-limb rehabilitation in adults with tetraplegia caused by cervical spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of traumatic incomplete (AIS B-D) cervical spinal cord injury (C8 and above)
* at least 12 months post-traumatic SCI but less than 10 years post-SCI
* demonstrate some residual movement in the upper limb (e.g., able to perform pinch movement with thumb and index finger sufficient to grip small objects such as marble)

Exclusion Criteria:

* non-traumatic SCI
* recent ear trauma and skin lesions at the site of stimulation, such as sunburn, cuts, and open sores,
* facial or ear pain,
* allergic reaction to adhesives and electrodes,
* any current or past history of cardiovascular disorders,
* intracranial metal implants, pacemakers,
* concomitant clinically significant brain injury,
* receiving medication that may significantly interfere with the actions of VNS on neurotransmitter systems at study entry
* If there is a plan for alteration in upper-extremity therapy or medication for muscle tone during the course of the study;
* medical or mental instability;
* pregnancy or plans to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of subjects with change in systolic blood pressure | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of subjects with change in diastolic blood pressure | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of subjects with change in heart rate | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of subjects with change in respiratory rate | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of subjects with change in autonomic dysreflexia | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of subjects with worsening spasticity | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of subjects with change in pain at stimulation site | Immediately after completing in-clinic 18 sessions (6-8 weeks)
Safety as assessed by number of adverse events that occurred during the study period | post therapy 30 days
Feasibility as assessed by the number of treatment sessions attended by each participant . The intervention is considered feasible if at least 80% adherence rate is achieved and no serious adverse events occurred. | from baseline through completion of 18 sessions (about 6-8 weeks)
  80% adherence rate is defined as completing ≥ 16 out of 18 sessions
Feasibility as assessed by the participants' perceptions of the study procedures | from baseline through completion of 18 sessions (about 6-8 weeks)
  This includes implementation using the paired taVNS with rehabilitation. This is numerically rated from 'not difficult at all' at 0, and 'very difficult' at 10, higher score indicating worse outcome
Feasibility as assessed by the participants' perceptions of the usefulness of the intervention | from baseline through completion of 18 sessions (about 6-8 weeks)
  This is numerically rated from ''not at all useful' at 0 and 'very useful' at 10 , higher score indicating better outcome

SECONDARY OUTCOMES:
Change in degree of upper limb impairment as assessed by the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) assessment | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  The 3 measured domains are as follows:
  1. Strength: Motor grading of 10 arm and hand muscles for right and left arm will be performed. Each muscle is graded from 0 to 5 for a maximum score of 50, a higher number indicating more strength.
  2. Dorsal and palmar sensation: Each test location is scored from 0 to 4. Three locations for the dorsal side of each hand and 3 for palmer location of each hand are summed to render a subtest total score between 0 and 12 a higher score indicating more sensation.
  3. Prehension:
     1. Qualitative prehension: The participant performs 3 tasks using each hand and is scored from 0-12 a higher number indicating a better outcome
     2. Quantitative prehension: he participant performs 6 tasks using each hand and is scored from 0-30 a higher number indicating a better outcome
Change in hand function as assessed by the Toronto Rehab Institute Hand Function Test (TRI-HFT) | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  This is a 14 item questionnaire and each is scored from 1(no movement elicited) to 8(normal grasp) a higher number indicating better hand function
Change in capability of using arms and hands as assessed by the Capabilities of Upper Extremity Questionnaire (CUE-Q) | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  This is a 17 item questionnaire and each is scored from 1(totally limited) to 7(not at all limited), a higher number indicating better outcome
Change in self care independence as assessed by the Spinal Cord Injury Independence Measure-III (SCIM-III) self-care subscore | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  This is a 4 item questionnaire and each is scored from 0(need total assistance) to 3(completely independent), higher score indicating more independence.
Change in Quality of Life as assessed by the Spinal Cord Injury- Quality of Life (SCI-QoL) questionnaire | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  This questionnaire has 3 parts:
  basic mobility: this is a 11 item questionnaire and each is scored from 1(unable to do) to 5(can do without difficulty)higher score indicating more mobility Fine Motor: This is a 9 item questionnaire and each is scored from 1(unable to do) to 5(can do without difficulty)higher score indicating better outcome self care: This is a 11 item questionnaire and each is scored from 1(unable to do) to 5(can do without difficulty)higher score indicating better outcome
Change in Pain as assessed by the International SCI pain basic data subset (version 2) | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  This is an 6 item questionnaire and each is scored from 0 (no pain) -10 (pain as bad as you can imagine), a higher score indicating more pain.
Change in Depression as assessed by the Patient Health Questionnaire (PHQ-8) | Baseline, immediately after completing in-clinic 18 sessions (6-8 weeks), post- therapy 30 days, and posttherapy 90 days]
  This is an eight item questionnaire and each is scored from 0(not at all) to 3(nearly every day) a higher score indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Radha Korupolu, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Neurorecovery Research Center, TIRR MHH, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No